CLINICAL TRIAL: NCT00540163
Title: Improvement in Physical Functioning (SF-36 Activity Score) in COPD Patients With Exercise-induced Dyspnoea on Treatment With Spiriva® 18 Microgram (Capsules Containing 18 μg Tiotropium).
Brief Title: Observational Non-interventional Study With Spiriva in Chronic Obstructive Pulmonary Disease Patients With Exercise-induced Dyspnoea
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.402
Record Dates: First submitted 2007-09-21; First posted 2007-10-05 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This observational non-interventional study is designed to demonstrate the improvement of physical function in COPD patients with exercise-induced dyspnoea on treatment with Spiriva (tiotropium 18 µg capsules) and allows adverse events to be recorded and evaluated.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion Criteria:

Men or women with COPD and a thoracic gas volume (TGV) of < 140% at rest, MRC value of 2 or more.

Exclusion Criteria:

* Patients cannot be recruited if any of the general or specific contraindications listed in the Patient information leaflet or the Summary of Product Characteristics applies.
* Tiotropium bromide inhalation powder is contraindicated in patients with a hypersensitivity to tiotropium bromide, atropine or its derivatives, e.g. ipratropium or oxitropium or to the excipient lactose monohydrate which contains milk protein.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of office-based pulmonology practices
Sampling Method: Probability Sample
Enrollment: 1296 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the proportion of patients with an improvement by ≥10 points in the standardised PF-10 score after 6 weeks of treatment with Spiriva® 18 Microgram | 6 weeks

SECONDARY OUTCOMES:
The secondary endpoint was the change in the standardised PF-10 score within 6 weeks of treatment with Spiriva® 18 Microgram | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (177):
- Germany (177):
  - Boehringer Ingelheim Investigational Site, Amberg
  - Boehringer Ingelheim Investigational Site, Anklam
  - Boehringer Ingelheim Investigational Site, Aschau
  - Boehringer Ingelheim Investigational Site, Auerbach
  - Boehringer Ingelheim Investigational Site, Augsburg
  - Boehringer Ingelheim Investigational Site, Backnang
  - Boehringer Ingelheim Investigational Site, Bad Doberan
  - Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site, Bad Oeynhausen
  - Boehringer Ingelheim Investigational Site, Bad Soden
  - Boehringer Ingelheim Investigational Site, Bad Wörishofen
  - Boehringer Ingelheim Investigational Site, Beelitz
  - Boehringer Ingelheim Investigational Site, Bensheim
  - Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Biberach
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site, Breisach
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Bruchsal
  - Boehringer Ingelheim Investigational Site, Buchholz
  - Boehringer Ingelheim Investigational Site, Bünde
  - Boehringer Ingelheim Investigational Site, Calw
  - Boehringer Ingelheim Investigational Site, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site, Celle
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - Boehringer Ingelheim Investigational Site, Coburg
  - Boehringer Ingelheim Investigational Site, Cologne
  - Boehringer Ingelheim Investigational Site, Cottbus
  - Boehringer Ingelheim Investigational Site, Darmstadt
  - Boehringer Ingelheim Investigational Site, Dillenburg
  - Boehringer Ingelheim Investigational Site, Dinslaken
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site, Düren
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site, Emden
  - Boehringer Ingelheim Investigational Site, Erbach im Odenwald
  - Boehringer Ingelheim Investigational Site, Erfurt
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Euskirchen
  - Boehringer Ingelheim Investigational Site, Fellbach
  - Boehringer Ingelheim Investigational Site, Flensburg
  - Boehringer Ingelheim Investigational Site, Forchheim
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Freising
  - Boehringer Ingelheim Investigational Site, Fürstenfeldbruck
  - Boehringer Ingelheim Investigational Site, Fürth
  - Boehringer Ingelheim Investigational Site, Gadebusch
  - Boehringer Ingelheim Investigational Site, Geilenkirchen
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Giessen
  - Boehringer Ingelheim Investigational Site, Gifhorn
  - Boehringer Ingelheim Investigational Site, Gotha
  - Boehringer Ingelheim Investigational Site, Göppingen
  - Boehringer Ingelheim Investigational Site, Greiz
  - Boehringer Ingelheim Investigational Site, Gummersbach
  - Boehringer Ingelheim Investigational Site, Gütersloh
  - Boehringer Ingelheim Investigational Site, Halberstadt
  - Boehringer Ingelheim Investigational Site, Halle
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamelin
  - Boehringer Ingelheim Investigational Site, Hamm
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Heilbronn
  - Boehringer Ingelheim Investigational Site, Herne
  - Boehringer Ingelheim Investigational Site, Hilden
  - Boehringer Ingelheim Investigational Site, Hildesheim
  - Boehringer Ingelheim Investigational Site, Hoyerswerda
  - Boehringer Ingelheim Investigational Site, Ibbenbueren
  - Boehringer Ingelheim Investigational Site, Ingolstadt
  - Boehringer Ingelheim Investigational Site, Iserlohn
  - Boehringer Ingelheim Investigational Site, Kaiserslautern
  - Boehringer Ingelheim Investigational Site, Kamen
  - Boehringer Ingelheim Investigational Site, Karlsruhe
  - Boehringer Ingelheim Investigational Site, Kaufbeuren
  - Boehringer Ingelheim Investigational Site, Kempten
  - Boehringer Ingelheim Investigational Site, Kevelaer
  - Boehringer Ingelheim Investigational Site, Kiel
  - Boehringer Ingelheim Investigational Site, Konstanz
  - Boehringer Ingelheim Investigational Site, Krefeld
  - Boehringer Ingelheim Investigational Site, Landshut
  - Boehringer Ingelheim Investigational Site, Langenfeld
  - Boehringer Ingelheim Investigational Site, Leipzig
  - Boehringer Ingelheim Investigational Site, Limburg
  - Boehringer Ingelheim Investigational Site, Lindenberg
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Lippstadt
  - Boehringer Ingelheim Investigational Site, Loerrach
  - Boehringer Ingelheim Investigational Site, Ludwigsburg
  - Boehringer Ingelheim Investigational Site, Lüdenscheid
  - Boehringer Ingelheim Investigational Site, Lüneburg
  - Boehringer Ingelheim Investigational Site, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, Marburg
  - Boehringer Ingelheim Investigational Site, Markkleeberg
  - Boehringer Ingelheim Investigational Site, Memmingen
  - Boehringer Ingelheim Investigational Site, Menden
  - Boehringer Ingelheim Investigational Site, Minden
  - Boehringer Ingelheim Investigational Site, Moers
  - Boehringer Ingelheim Investigational Site, Mönchengladbach
  - Boehringer Ingelheim Investigational Site, Mühldorf
  - Boehringer Ingelheim Investigational Site, Mülheim
  - Boehringer Ingelheim Investigational Site, München
  - Boehringer Ingelheim Investigational Site, Neu-Ulm
  - Boehringer Ingelheim Investigational Site, Neunkirchen
  - Boehringer Ingelheim Investigational Site, Norderstedt
  - Boehringer Ingelheim Investigational Site, Nordhausen
  - Boehringer Ingelheim Investigational Site, Nuremberg
  - Boehringer Ingelheim Investigational Site, Oberursel
  - Boehringer Ingelheim Investigational Site, Olpe
  - Boehringer Ingelheim Investigational Site, Oschersleben
  - Boehringer Ingelheim Investigational Site, Osnabrück
  - Boehringer Ingelheim Investigational Site, Papenburg
  - Boehringer Ingelheim Investigational Site, Peine
  - Boehringer Ingelheim Investigational Site, Plauen
  - Boehringer Ingelheim Investigational Site, Potsdam
  - Boehringer Ingelheim Investigational Site, Pulheim
  - Boehringer Ingelheim Investigational Site, Rastatt
  - Boehringer Ingelheim Investigational Site, Rathenow
  - Boehringer Ingelheim Investigational Site, Regensburg
  - Boehringer Ingelheim Investigational Site, Remscheid
  - Boehringer Ingelheim Investigational Site, Rendsburg
  - Boehringer Ingelheim Investigational Site, Rostock
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
  - Boehringer Ingelheim Investigational Site, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site, Saarbrücken
  - Boehringer Ingelheim Investigational Site, Saarlouis
  - Boehringer Ingelheim Investigational Site, Salzgitter
  - Boehringer Ingelheim Investigational Site, Schenefeld
  - Boehringer Ingelheim Investigational Site, Schleswig
  - Boehringer Ingelheim Investigational Site, Schmölln
  - Boehringer Ingelheim Investigational Site, Schwalmstadt
  - Boehringer Ingelheim Investigational Site, Schwalmtal
  - Boehringer Ingelheim Investigational Site, Schwerin
  - Boehringer Ingelheim Investigational Site, Sebnitz
  - Boehringer Ingelheim Investigational Site, Seevetal
  - Boehringer Ingelheim Investigational Site, Siegen
  - Boehringer Ingelheim Investigational Site, Singen
  - Boehringer Ingelheim Investigational Site, Sinsheim
  - Boehringer Ingelheim Investigational Site, Solingen
  - Boehringer Ingelheim Investigational Site, Sonneberg
  - Boehringer Ingelheim Investigational Site, Spremberg
  - Boehringer Ingelheim Investigational Site, Stade
  - Boehringer Ingelheim Investigational Site, Starnberg
  - Boehringer Ingelheim Investigational Site, Steinbach
  - Boehringer Ingelheim Investigational Site, Straelen
  - Boehringer Ingelheim Investigational Site, Strausberg
  - Boehringer Ingelheim Investigational Site, Stuttgart
  - Boehringer Ingelheim Investigational Site, Teltow
  - Boehringer Ingelheim Investigational Site, Teterow
  - Boehringer Ingelheim Investigational Site, Troisdorf
  - Boehringer Ingelheim Investigational Site, Unna
  - Boehringer Ingelheim Investigational Site, Uttenreuth
  - Boehringer Ingelheim Investigational Site, Verden an der Aller
  - Boehringer Ingelheim Investigational Site, Waiblingen
  - Boehringer Ingelheim Investigational Site, Waren
  - Boehringer Ingelheim Investigational Site, Warendorf
  - Boehringer Ingelheim Investigational Site, Weiden
  - Boehringer Ingelheim Investigational Site, Weißenhorn
  - Boehringer Ingelheim Investigational Site, Wetzlar
  - Boehringer Ingelheim Investigational Site, Wiesloch
  - Boehringer Ingelheim Investigational Site, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site, Witten
  - Boehringer Ingelheim Investigational Site, Worms
  - Boehringer Ingelheim Investigational Site, Wuppertal
  - Boehringer Ingelheim Investigational Site, Zella-Mehlis
  - Boehringer Ingelheim Investigational Site, Zossen